CLINICAL TRIAL: NCT07354035
Title: A Prospective, Randomized, Multicenter Clinical Trial in Evaluating the Safety and Efficacy of the Use of Coronary Sinus Balloon Pump Along With PCI in STEMI Patients
Brief Title: The Coronary Sinus Balloon Pump in STEMI
Acronym: REVIVE-RCT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai MicroPort Rhythm MedTech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AMD-D-005
Record Dates: First submitted 2026-01-05; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: STEMI
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The coronary sinus balloon pump +PCI (Experimental): Subjects in the experimental group will be treated with the coronary sinus balloon pump manufactured by Shanghai Microport Rotapace Co. Ltd.
  Interventions: Device: The coronary sinus balloon pump; Procedure: Percutaneous Coronary Intervention (PCI)
- Standard PCI (Placebo Comparator)
  Interventions: Procedure: Percutaneous Coronary Intervention (PCI)

INTERVENTIONS:
Device: The coronary sinus balloon pump — The coronary sinus balloon pump comprises a coronary sinus balloon pump catheter system and a coronary sinus balloon pump therapeutic device. This product is indicated for the treatment of ST-segment elevation myocardial infarction (STEMI) with or without coronary microvascular dysfunction (CMD), by intermittently occluding coronary sinus blood flow during percutaneous coronary intervention (PCI) procedures to reduce myocardial infarction size.
  Arms: The coronary sinus balloon pump +PCI
Procedure: Percutaneous Coronary Intervention (PCI) — Minimally invasive procedures used to open clogged coronary arteries

SUMMARY:
This study is a prospective, multicenter, randomized controlled clinical trial designed to evaluate the safety and efficacy of the coronary sinus balloon pump (manufactured by Shanghai MicroPort Rotapace Medical Technology Co., Ltd.) as an adjunctive therapy during percutaneous coronary intervention (PCI) in patients with acute ST-segment elevation myocardial infarction (STEMI). As a pivotal study, it aims to support the product registration application to the National Medical Products Administration (NMPA).

ELIGIBILITY:
Inclusion Criteria:

General Inclusion Criteria:

1. Subjects aged ≥18 and ≤80 years, clinically diagnosed with ST-segment elevation myocardial infarction (STEMI).
2. Left ventricular ejection fraction (LVEF) ≤50% and ≥35% as assessed by echocardiography or left ventriculography prior to PCI.
3. Symptoms of myocardial infarction (e.g., persistent chest pain, with or without shortness of breath, nausea/vomiting, profuse sweating, dyspnea, syncope) consistent with the timing of myocardial ischemia, with symptom onset within 24 hours.
4. Electrocardiographic evidence of acute anterior wall myocardial infarction, defined as ST-segment elevation ≥1 mm (0.1 mV) in at least two contiguous precordial leads on a 12-lead ECG. For leads V2 or V3, the following gender- and age-specific cutoffs apply:

   * 2 mm (0.2 mV) in men ≥45 years old.
   * 2.5 mm (0.25 mV) in men <40 years old.
   * 1.5 mm (0.15 mV) in women.
5. Subject is eligible for primary percutaneous coronary intervention (primary PCI).
6. Subject is able to understand the purpose of the study, voluntarily agrees to participate by signing the informed consent form acknowledging the risks and benefits described therein, and is willing and able to comply with the required clinical follow-up procedures.

Angiographic Inclusion Criteria:

1. The target lesion is located in the proximal or mid segment of the left anterior descending artery (LAD).
2. TIMI flow grade of the target vessel is 0, 1, or 2 prior to PCI treatment.

Exclusion Criteria:

1. Presence of an implant or foreign body within the coronary sinus.
2. The target lesion involves the left main coronary artery, or there is a ≥50% stenosis in the left main coronary artery.
3. Known allergy or contraindication to drugs or materials required during PCI and the use of the investigational device (including, but not limited to, sirolimus, dual antiplatelet therapy drugs, polyamide, polyurethane, polytetrafluoroethylene, or stainless steel).
4. Presence of pericardial effusion (moderate or greater), cardiac tamponade, hemodynamically significant left/right shunt, or severe valvular heart disease.
5. Intracardiac thrombus detected by echocardiography within 30 days prior to enrollment.
6. History of acute myocardial infarction, or documented history of hospitalization for Q-wave infarction.
7. History of cerebral infarction, intracerebral hemorrhage, transient ischemic attack (TIA), or reversible ischemic neurologic deficit within the past 6 months, or presence of permanent neurological deficit.
8. Known hemoglobin level below 90 g/L, platelet count below 80×10⁹/L, history of bleeding diathesis or coagulation disorder, or unwillingness to receive blood transfusion.
9. Subjects requiring circulatory support or assisted ventilation.
10. Subjects experiencing cardiac arrest or cardiopulmonary resuscitation (CPR) for more than 5 minutes preoperatively (baseline) or intraoperatively.
11. Subjects unsuitable for femoral or jugular venous access.
12. Known contraindications to cardiac magnetic resonance imaging (CMR), such as claustrophobia, presence of non-CMR compatible foreign bodies or implants, or allergy/intolerance to gadolinium-based contrast agents.
13. Prior coronary artery bypass graft (CABG) surgery.
14. Visible well-developed collateral circulation distal to the target lesion in the target vessel.
15. Current participation in another clinical drug or device study where the primary endpoint has not been reached, or planned participation in another investigational drug or device clinical trial within 12 months after the baseline procedure.
16. Known severe renal disease (estimated glomerular filtration rate (eGFR) <30 mL/(min·1.73m²) as calculated by the MDRD formula*) or undergoing hemodialysis.
17. History of treatment for malignancy within the past 12 months.
18. Subjects with chronic obstructive pulmonary disease (COPD) who are on home oxygen therapy or receiving chronic steroid therapy.
19. Impaired consciousness during PCI, cardiogenic shock (persistent systolic blood pressure ≤90 mmHg despite conservative treatment), or pulmonary edema (peripheral oxygen saturation <90% with rales).
20. Any vascular PCI treatment received within 1 week prior to enrollment.
21. Fibrinolytic therapy received within 24 hours prior to enrollment.
22. -target lesions in vessels other than the left anterior descending artery and its branches requiring treatment during this PCI or within one week thereafter.
23. Known pregnancy or breastfeeding, or female subjects planning pregnancy within 1 year post-procedure and unable to complete follow-up as required.
24. Subjects judged by the investigator to have poor compliance and unable to complete the study as required, or any other reason the investigator deems the subject unsuitable for enrollment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 177 (Estimated)
Dates: Start 2026-02-12 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Myocardial infarct size | 5 days after the procedure
  Myocardial infarct size is measured by cardiac magnetic resonance (CMR) 5 days after the procedure, expressed as a percentage of left ventricular mass (%LV).
Incidence of Major Adverse Events (MAE) (Experimental Group) | at 30 days post-procedure
  Major Adverse Events (MAE) include:
  All-cause death Myocardial infarction Target vessel revascularization Hospitalization for heart failure New onset or worsening heart failure Coronary sinus dissection or perforation requiring intervention or surgical repair Thrombosis or thromboembolism Stroke Major bleeding (BARC Type 3~5) Ventricular tachycardia or ventricular fibrillation requiring defibrillation or cardioversion

SECONDARY OUTCOMES:
Device Success Rate (Experimental Group) | Immediately post-procedure
  Successful delivery and deployment of the device to the coronary sinus and completion of the intended procedure
Procedure Success Rate (Experimental Group) | Immediately post-procedure
  Achievement of PCI success based on device success, without the occurrence of any CSBP-related adverse events
Coronary Sinus Pressure (Experimental Group) | Immediately post-procedure
Change in ST-Segment Elevation | Immediately post-procedure
  Change in ST-Segment Elevation [Comparison between post-PCI ECG and baseline]
Incidence of Device-Related Procedural Complications (Experimental Group) | Immediately post-procedure
  Procedural Complications are defined as: Access site complications (including access site bleeding of BARC Type 3-5, access site infection requiring oral or intravenous antibiotics, access site complication requiring surgical intervention), coronary sinus dissection or perforation requiring intervention or surgical repair, pericardial effusion or cardiac tamponade requiring intervention or surgical treatment, thrombosis or thromboembolism, and stroke. The relatedness of a procedural complication to the device must be adjudicated by the Clinical Events Committee (CEC).
Death (cardiac, vascular, non-vascular) | at 5 days, 30 days, 6 months, and 12 months post-procedure
  Rate of death (cardiac, vascular, non-vascular), as adjudicated by the Clinical Events Committee (CEC)
Rate of heart failure hospitalization | at 5 days, 30 days, 6 months, and 12 months post-procedure
Incidence of new-onset or worsening heart failure | at 5 days, 30 days, 6 months, and 12 months post-procedure
Incidence of myocardial infarction | at 5 days, 30 days, 6 months, and 12 months post-procedure
Incidence of revascularization (target lesion, target vessel, any coronary) | at 5 days, 30 days, 6 months, and 12 months post-procedure
Incidence of stent thrombosis | at 5 days, 30 days, 6 months, and 12 months post-procedure
Incidence of major bleeding events | at 5 days, 30 days, 6 months, and 12 months post-procedure
Incidence of stroke | at 5 days, 30 days, 6 months, and 12 months post-procedure
Severity of angina | at 5 days, 30 days, 6 months, and 12 months post-procedure
  Angina severity (classified according to the Canadian Cardiovascular Society Classification of Angina Pectoris) is assessed by the level of physical activity that triggers the chest pain. And the lower the level that triggers the chest pain, the more serious angina.
Ventricular tachycardia or ventricular fibrillation requiring defibrillation or cardioversion | at 5 days, 30 days, 6 months, and 12 months post-procedure
  Ventricular tachycardia or ventricular fibrillation requiring defibrillation or cardioversion as adjudicated by the CEC
EQ-5D quality of life score | at 5 days, 30 days, 6 months, and 12 months post-procedure
  Changes in quality of life measured by EQ-5D (assessed by the following five dimensions: mobility, self-care, usual activities, pain/discomfort, anxiety/depression) (scale of 0-100: higher score better)
Incidence of adverse events and serious adverse events | at 5 days, 30 days, 6 months, and 12 months post-procedure
Incidence of device deficiencies (Experimental Group only) | at 5 days, 30 days, 6 months, and 12 months post-procedure